CLINICAL TRIAL: NCT06439381
Title: A Multicenter, Randomized, Continuing Trial to Evaluate the Long-term Safety and Efficacy of TQH2722 Injection in the Treatment of Chronic Sinusitis With or Without Nasal Polyps
Brief Title: Long-term Safety and Efficacy of TQH2722 Injection in the Treatment of Chronic Sinusitis With or Without Nasal Polyps
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQH2722-II-04
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2023-11

CONDITIONS: Chronic Rhinosinusitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 300mg/600mg of TQH2722 injection in Part A or B (Experimental): For Part A or Part B, 300mg/600mg of TQH2722 injection was administered every 2 weeks until week 22, combined with Mometasone furoate nasal spray of 100-200μg/ day until week 32.
  Interventions: Drug: 300mg/600mg of TQH2722 injection

INTERVENTIONS:
Drug: 300mg/600mg of TQH2722 injection — TQH2722 injection is a fully human monoclonal antibody that interfering with the signal cascade.

SUMMARY:
This is a multicenter, randomized, continuing, Phase II expansion trial to evaluate the safety, efficacy, and immunogenicity of two doses of TQH2722 in the long-term treatment of severe chronic sinusitis with or without nasal polyps.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion Criteria of Part A

   * Sign informed consent before the test to fully understand the purpose, process and possible adverse reactions of the test;
   * Age 18-75 years old (including the threshold), male or female;
   * Enroll in the clinical study of TQH2722 for chronic sinusitis with or without nasal polyps (study number TQH2722-II-02) and meet the following criteria "a" or "b" :

     1. Subjects completed prescribed treatment as required and completed Part A end of study (EOS) visit;
     2. The subjects withdrew early due to poor compliance or other objective reasons other than TQH2722-related AE, and completed the early exit interview according to the plan, and the influencing factors that led to the subjects' early termination of the main study treatment have disappeared/no longer affected the subjects' participation in the continuation study as assessed by the investigators and sponsors.

   Note: If protocol window period requirements are met, examination results from subject's main study EOS/ early exit visit may be used as screening/baseline examination for this study.
   * Subjects had used a more stable dose of nasal glucocorticoids (INCS) for more than 4 weeks prior to screening (for subjects who had used other INCS prior to screening than intranasal Mometasone furoate nasal spray (MFNS), subjects were willing to switch to MFNS during the study);
   * Subjects agree not to have a family plan for 6 months from the date of signing the informed consent to the last dose, and must use effective non-drug contraception with their sexual partners of childbearing age.
2. Inclusion Criteria of Part B

   * Sign informed consent before the test to fully understand the purpose, process and possible adverse reactions of the test;
   * Age 18-75 years old (including the threshold), male or female;
   * Enroll in the clinical study of TQH2722 for chronic sinusitis with or without nasal polyps (study number TQH2722-II-02) and meet the following criteria "a" or "b" :

     1. Subjects completed prescribed treatment as required and completed Part B EOS visit;
     2. The subjects withdrew early due to poor compliance or other objective reasons other than TQH2722-related AE, and completed the early exit interview according to the plan, and the influencing factors that led to the subjects' early termination of the main study treatment have disappeared/no longer affected the subjects' participation in the continuation study as assessed by the investigators and sponsors.

Note: If protocol window period requirements are met, examination results from subject's main study EOS/ early exit visit may be used as screening/baseline examination for this study.

* Subjects had used a more stable dose of nasal glucocorticoids (INCS) for more than 4 weeks prior to screening (for subjects who had used other INCS prior to screening than intranasal Mometasone furoate nasal spray (MFNS), subjects were willing to switch to MFNS during the study);
* Subjects agree not to have a family plan for 6 months from the date of signing the informed consent to the last dose, and must use effective non-drug contraception with their sexual partners of childbearing age.

Exclusion Criteria:

* In the main study (TQH2722-II-02), a TQH2722-related SAE occurred or TQH2722-related AE led to the discontinuation of TQH2722 therapy, and after discussion between the investigator and sponsor, the subject was deemed unsuitable for continuation of TQH2722 therapy.
* The subjects had poor compliance in the main study, and the researchers judged that they could not complete the continuing study.
* During the main study (TQH2722-II-02), any severe progression or poorly controlled concomitant disease (such as asthma exacerbation requiring adjustment of background medication) is identified and the subject is deemed unfit to participate by the principal investigator;
* Any of the following laboratory test values are abnormal during the screening period:

  1. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2.5 upper limit of normal (ULN);
  2. Total bilirubin > 2 x ULN (except indirect bilirubin elevation secondary to Gilbert syndrome);
  3. Creatinine > 1.5×ULN;
* Any medical condition, including but not limited to cardiovascular, gastrointestinal, liver, kidney, neurological, musculoskeletal, infectious, endocrine, metabolic, hematological, psychiatric, or major limb disorders, that the investigator believes is unstable and may affect the patient's safety throughout the study period, or affect the study results or their interpretation, or interfere with the patient's ability to complete the entire study process.For example, but not limited to: ischemic heart disease, left ventricular failure, arrhythmia, uncontrolled hypertension, uncontrolled hyperglycemia, cerebrovascular disease, etc.;
* Patients with active autoimmune diseases (including, but not limited to, Hashimoto thyroiditis, Graves' disease, inflammatory bowel disease, primary biliary cholangitis, systemic lupus erythematosus, multiple sclerosis and other neuroinflammatory diseases, psoriasis vulgaris, rheumatoid arthritis);
* Known or suspected immunosuppressed individuals, including but not limited to a history of invasive opportunistic infections (e.g., histoplasmosis, listeriosis, coccidioidomycosis, pulmonary cyst disease, aspergillosis), even if the infection has resolved;
* Subjects with active malignant tumors or a history of malignant tumors:Patients with basal cell carcinoma, skin localized squamous cell carcinoma, or cervical carcinoma in situ who had completed curative treatment for at least 12 months prior to visit 1 could be enrolled in this study; patients with other malignancies could be enrolled if they had completed curative treatment for at least 5 years prior to visit 1;
* A history of active pulmonary tuberculosis within 12 months prior to screening;
* Active hepatitis was present at the screening stage, either hepatitis B surface antigen (HBsAg) positive, hepatitis B core antibody (HBcAb) positive and Hepatitis B Virus-DNA positive, or Hepatitis C Virus (HCV) antibody positive and HCV-RNA positive; or human immunodeficiency virus (Anti-HIV) positive, or treponema pallidum antibody (Anti-TP) positive (if the treponema pallidum serological test is positive, then further non-treponema pallidum serological test is performed, the latter is negative and the investigator determines that patients who have been infected with syphilis in the past but have been cured are eligible for inclusion);
* Diagnosis of helminthic infection within 6 months prior to the screening period, failure to receive standard treatment or failure to respond to standard treatment;
* Subjects who received the following treatments:

  1. Had sinus surgery or nasal sinus surgery within 6 months prior to screening (visit 1).
  2. Received monoclonal antibody therapy within 8 weeks or 5 half-lives prior to screening (whichever is longer);
  3. Received immunosuppressive therapy (including but not limited to cyclophosphamide, cyclosporine, interferon gamma, azathioprine, methotrexate, mycophenolate and tacrolimus) within 8 weeks or 5 half-lives prior to screening, whichever is longer;
  4. Use of other non-biological agents within 8 weeks or 5 half-lives (whichever is longer) prior to screening;
  5. Intravenous immunoglobulin (IVIG) therapy and/or plasma exchange within 30 days prior to screening visit (Visit 1);
  6. Subjects treated with leukotriene antagonists/modulators prior to screening (subjects treated with stable doses of leukotriene modulators for ≥30 days prior to screening can be enrolled);
  7. Start allergen immunotherapy within 3 months prior to screening, or plan to start such therapy during the study period or plan to change the therapeutic dose during the study period;
  8. Have received live attenuated vaccine within 4 weeks prior to screening or plan to receive live attenuated vaccine during the study period;
  9. Chronic active or acute infection requiring systemic treatment with antibiotics, antivirals, antiparasites, antivirals, or antifungals during the 4 weeks prior to screening, or a viral disease that may not have received antiviral treatment during the 4 weeks prior to screening;(Screening visits can be performed after the patient recovers from infection, but the systemic antibiotic washout period needs to be greater than 2 weeks).
* Patients with asthma should be excluded if: a. forced expiratory volume in the first second (FEV1) ≤ 50% of the expected normal value, or b.Acute exacerbation of asthma within 90 days prior to screening requiring hospitalization (>24 hours), or c.Are using a daily dose of fluticasone or equivalent inhaled glucocorticoids (ICS) greater than 1000mcg;
* Subjects with asthma were initiated with inhaled corticosteroids within 4 weeks prior to the screening/induction period (for subjects who could receive a stable dose for at least 4 weeks prior to screening and whose assessed dose could be maintained throughout the study period, inhaled corticosteroids could be fluticasone propionate at a dose ≤1000μg or equivalent doses of other inhaled corticosteroids).
* Subjects have concomitant medical conditions that prevent them from completing the screening period assessment or evaluating the primary efficacy endpoint, such as:

  1. A deviated nasal septum leads to obstruction of at least one nostril
  2. Persistent drug rhinitis;
  3. The diagnosis was eosinophilic granulomatous vasculitis (Churg-Strauss syndrome), granulomatous polyvasculitis (Wegener's granuloma), Young's syndrome, Kartagener syndrome or other ciliary dyskinesia syndrome, cystic fibrosis;
  4. Suspected or confirmed fungal rhinosinusitis on imaging;
* Subjects with nasal malignancies and benign tumors (e.g., papilloma, hemangioma, etc.);
* Subjects who are unable to use MFNS or are allergic or intolerant to Mometasone furoate nasal spray;
* Subjects with a history of systemic allergy to any biological agent (except local injection site reactions);
* Pregnant or lactating women;
* Alcohol, drug and known drug dependence;
* The subjects had poor compliance in the study and could not complete the study as judged by the researcher;
* Any medical or psychiatric condition that, in the judgment of the investigator or sponsor medical reviewer, puts the subject at risk, interferes with participation in the study, or interferes with the interpretation of the study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-07-16 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Treatment emergent adverse events (TEAE) | Up to 32 weeks
  Frequency of treatment emergent adverse events (TEAE) occurring during treatment.

SECONDARY OUTCOMES:
Serious adverse events (SAEs) | Up to 32 weeks
  The frequency of serious adverse events (SAEs) that occurred during treatment in subjects with chronic sinusitis with nasal polyps (CRSwNP) or chronic sinusitis without nasal polyps (CRSsNP).
Abnormal laboratory test indicators | Up to 32 weeks
  Abnormal laboratory test indicators during treatment in subjects with chronic sinusitis with nasal polyps (CRSwNP) or chronic sinusitis without nasal polyps (CRSsNP).
Changes in Lund Mackay score assessed by CT from baseline | Up to 24 weeks
  Change in Lund Mackay score assessed by CT from baseline. The total score is 0-24 points, with the higher score meaning the more severe symptoms.
Changes in the University of Pennsylvania Smell Identification Test (UPSIT) | Up to 32 weeks
  The change in the University of Pennsylvania Smell Identification Test (UPSIT) from baseline (main study TQH2722-II-02 and baseline in this study, respectively) at each evaluation time point.
Changes in Nasal Total Symptom Score from baseline | Up to 32 weeks
  Changes in subjects' Nasal Total Symptom Score from baseline. The total score is 0-9 points, with the higher score meaning the more severe symptoms.
Changes in the sinusitis Visual Analogue Scale (VAS) score from baseline | Up to 32 weeks
  Changes in the sinusitis Visual Analogue Scale (VAS) score from baseline were measured at each evaluation time point. The total score is 0-10 points, with the higher score meaning the more severe symptoms.
Immunogenicity: The incidence of drug-resistant antibodies (ADA) and their titers, and the incidence of neutralizing antibodies (Nab). | 0h (The first dose), D113, D169 and during withdrawal
  Immunogenicity: The incidence of drug-resistant antibodies (ADA) and their titers, and the incidence of neutralizing antibodies (Nab) in subject. If the subject tests positive for ADA, neutralizing antibodies are added.
Changes in nasal polyp scores of subjects with chronic sinusitis with nasal polyps (CRSwNP) in part A | Weekends 0, 8, 16, 24 and 32
  Changes in nasal polyp scores of subjects with chronic sinusitis with nasal polyps (CRSwNP) at each evaluation time point were compared with baseline values (TQH2722-II-02 in the main study and baseline values in this study, respectively).
Changes in Sino-nasal Outcome Test (SNOT-22) in part A | Weekends 0, 8, 16, 24 and 32
  Changes in Sino-nasal Outcome Test (SNOT-22) from baseline for subjects at each evaluation time point.
Changes in nasal congestion score (NCS) in part A from baseline | Up to 32 weeks
  The changes in nasal congestion score (NCS) from baseline at each evaluation time point in Part A. The total score is 0-3 points, with the higher score meaning the more severe symptoms.
Changes in nasal/posterior runny nose scores in part A from baseline | Up to 32 weeks
  Changes in subjects' nasal/posterior runny nose scores from baseline at each evaluation time point. The total score is 0-3 points, with the higher score meaning the more severe symptoms.
Changes in the anosmia score in part A from baseline | Up to 32 weeks
  The changeS in the anosmia score from baseline at each evaluation time point in part A. The total score is 0-3 points, with the higher score meaning the more severe symptoms.
Changes of olfactory loss score in part B from baseline | Up to 32 weeks
  In Part B, the change of subjects' olfactory loss score from baseline (using the main study TQH2722-II-02 and the baseline value in this study, respectively) at each evaluation time point. The total score is 0-3 points, with the higher score meaning the more severe symptoms.
Changes in nasal endoscopic modified Lund-Kennedy scores in part B | Weekends 0, 8, 16, 24 and 32
  In Part B, changes in subjects' nasal endoscopic modified Lund-Kennedy scores from baseline (using the main study TQH2722-II-02 and the baseline in this study, respectively) at each evaluation time point are measured. The total score is 0-24 points, with the higher score meaning the more severe symptoms.
Changes in Sino-nasal Outcome Test (SNOT-22) in part B | Weekends 0, 8, 16, 24 and 32
  In Part B, change from baseline in Sino-nasal Outcome Test (SNOT-22) for subjects at each evaluation time point.

CONTACTS AND LOCATIONS:
Locations (27):
- China (27):
  - Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First People's Hospital of Foshan, Foshan, Guangdong
  - The Second People's Hospital of Shenzhen, Shenzhen, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Hebei Medical University Third Hospital, Shijiazhuang, Hebei
  - Cangzhou Central Hospital, Cangzhou, Heibei
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of science and technology, Wuhan, Hubei
  - Renmin Hospital of Wuhan University Hubei General Hospital, Wuhan, Hubei
  - Loudi Central Hospital, Changsha, Hunan
  - Baotou Central Hospital, Baotou, Inner Mongolia
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Jilin Provincial People's Hospital, Changchun, Jilin
  - The Affiliated Hospital of Yanbian University, Yanji, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Shengjing Hospital Affiliated to China Medical University, Shenyang, Liaoning
  - The Central Hospital of Shenyang Medical College, Shenyang, Liaoning
  - Shandong Second People's Hospital, Jinan, Shandong
  - Weihai Central Hospital, Weihai, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Zibo Central Hospital, Zibo, Shandong
  - Renji Hospital Shanghai Jiaotong University School of Medical, Shanghai, Shanghai Municipality
  - First Hospital of Shangxi Medical University, Taiyuan, Shangxi
  - Chengdu Second People's Hospital, Chengdu, Sichuan
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Taizhou central hospital(Taizhou university hospital), Taizhou, Zhejiang
  - Wenling First People's Hospital, Wenling, Zhejiang